CLINICAL TRIAL: NCT04038476
Title: Prospective, Randomised Evaluation of Transcutaneous Carbon-dioxide Monitoring in Complex Electrophysiological Procedures in Deep Sedation
Brief Title: Transcutaneous Carbon-dioxide Monitoring in Electrophysiological Procedures in Deep Sedation
Acronym: TRACES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Dr Karolina Weinmann, Cardiologist, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCM1
Record Dates: First submitted 2019-07-15; First posted 2019-07-30 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Conscious Sedation During Procedure; Ablation of Arrhythmias
Keywords: electrophysiology; conscious sedation; transcutaneous CO2 measurement; sedation monitoring; ablation of arrhythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard monitoring (Other): When assigned to the group "Standard monitoring":
  In the area of the forehead of the patient, the adhesive electrode is attached according to manufacturer's instructions before the first dose of sedatives. The sedation monitoring is performed under standard conditions by continuous measurement of oxygen saturation, continuous circulatory monitoring (heart rate and regular non-invasive blood pressure measurements) and half-hourly venous blood gas analysis, on receipt in the left atrium an additional arterial blood gas analysis. The examiner (doctor or physicians involved in the study) are blinded to the transcutaneous CO2 measurement. An adjustment of the sedation management therefore takes place on the basis of the monitoring measures mentioned above. Transcutaneous CO2 monitoring is recorded in the background (Excel table of all registered values) and also monitored by the sedation assisting nurse and integrated into the standard sedation protocol.
  Interventions: Diagnostic Test: Standard monitoring
- Standard monitoring + transcutaneous CO2 monitoring (Other): When assigned to the group "Standard monitoring + transcutaneous CO2 monitoring":
  In the area of the forehead of the patient, the adhesive electrode is attached according to manufacturer's instructions before the first dose of sedatives. The sedation monitoring is performed under standard conditions by continuous measurement of oxygen saturation, continuous circulatory monitoring (heart rate and regular non-invasive blood pressure measurements) and half-hourly venous blood gas analysis, on receipt in the left atrium an additional arterial blood gas analysis. In this group, the values of transcutaneous, continuous CO2 monitoring, including an alarm sound, are accessible to the treating physicians. Moreover, sedation management is adjusted on the basis of transcutaneous CO2 measurement. The above-mentioned measurements of the standard monitoring are carried out as described, in addition there is the the transcutaneous CO2 monitoring.
  Interventions: Diagnostic Test: Standard monitoring + transcutaneous CO2 monitoring

INTERVENTIONS:
Diagnostic Test: Standard monitoring + transcutaneous CO2 monitoring — The transcutaneous CO2 Monitoring measures the CO2 partial pressure of the skin and in condition of good circulation these values approximate the arterial/venous CO2 partial pressure. The sensor is placed on the forehead. The physician adapts the sedation Management according to the transcutaneous CO2 monitoring.
  Arms: Standard monitoring + transcutaneous CO2 monitoring
Diagnostic Test: Standard monitoring — The transcutaneous CO2-sensor is also positioned on the patients' forehead, but the transcutaneous CO2-monitoring is not available for the physician to adapt the sedative management.
  Arms: Standard monitoring

SUMMARY:
Complex procedures for treatment of cardiac arrhythmias are usually performed under deep sedation, since a quiet position of the patient is usually required over several hours and a significant risk of injury is caused by unconsciously movements of the patient. The sedative medication inhibits respiration. This can result in an increase of CO2-levels or a reduction oxygen-levels in the blood. Therefore, oxygen saturation (finger clip) is monitored continuously and the CO2-levels in the blood are evaluated every half hour. The study aims to evaluate, whether additional continuous CO2 measurement (transcutaneous CO2 monitoring) has a safety benefit for patients in sedation. Patients are randomly divided into two groups. The first group receives the previous standard monitoring and the second group additionally receives the transcutaneous CO2 measurement. After completion of the procedure, all study-relevant parameters are collected. Finally, the investigators examine whether oxygen saturation decreases or CO2-level increases could be prevented by a continuous, transcutaneous CO2 measurement.

DETAILED DESCRIPTION:
Complex catheter ablations for treatment of supraventricular and ventricular tachycardias are performed under moderate to deep sedation.

These interventions include electrophysiological examinations such as cryo-pulmonary vein isolation as well as complex radiofrequency ablation using a 3D mapping system. In order to avoid complications and to achieve a successful ablation result, a quiet position of the patient should be ensured during the examination, which usually lasts several hours. Specific reasons for the need for sedation include:

1. Femoral access The access is, in most cases, the right femoral vein. By transseptal puncture of the atrial septum, the catheters are inserted into the left atrium, the most common target structure of the above mentioned procedures. In order to insert the catheter safely into the left atrium, the path from the right groin to the left atrium is secured by a guide rail, a so-called sheath. Due to this relatively rigid guide rail, unconsciously movements of the patient should be avoided during the examination.
2. 3D mapping system The 3D mapping system is used to create an individual, virtual, electro-anatomical map ("map of the structure and electrical activity of the heart") of the left atrium of the patient. The prerequisite for a millimeter accurate determination of the catheter position by means of magnetic fields is the patient's quiet position. Already deep breaths can endanger the catheter stability and thus the ablation result. By movements of the patient there is also the risk that the virtual 3D map no longer matches the real anatomy, this results in an increased risk of perforation in the left heart with the result of a pericardial effusion or tamponade.
3. Patient positioning The patient has to lie flat and quiet during the procedure. Keeping this position presents a challenge even for younger patients and short examination times and is therefore impractical for the patient for several hours for reasons of comfort.

The sedation usually consists of a combination of midazolam and propofol. At the beginning of the study, a midazolam bolus is administered and a low-dose propofol perfusor is started, which is increased during the course until an optimal sedation depth is reached. During ablation, opiates are also added for analgesia, depending on the procedure, consisting of fentanyl single doses or continuous administration of remifentanil with perfusor.

The sedation depth is primarily controlled clinically. The above-mentioned substances all have a respiratory depressive effect and can cause respiratory complications, in the sense of hypercapnia or hypoxia. Therefore, standard monitoring involves the continuous measurement of oxygen saturation by means of pulse oximetry (spO2) as well as the half-hourly analysis of a venous blood gas analysis to evaluate the pH and to monitor the carbon dioxide partial pressure (pCO2). For interventions in the left atrium there is also the possibility of an arterial blood gas analysis from the left atrium or, if present, arterial blood gas analysis from an arterial sheath. If abnormalities occur in the blood gas analysis, the depth of sedation is adjusted accordingly or the dosage of the various components of the sedation is adapted. In addition, there is a continuous heart rate measurement and regular non-invasive blood pressure measurements. The nurse, assisting the sedation, also provides a dedicated sedation protocol, with explanations of any change in sedation management during the procedure.

In the electrophysiology laboratory of the ulm university hospital is the option of continuous, transcutaneous CO2 monitoring using TCM 400 (Radiometer). For this purpose, an adhesive electrode (Severinghaus electrode) is attached to the forehead of the patient. Hereby, the measurement of the O2 and CO2 partial pressure in the underlying tissue can take place and with good blood flow, this value approaches the invasively gained gas values. This method ensures a continuous, non-invasive CO2 measurement. The collected parameters are stored by the TCM 400 device in an Excel spreadsheet and can be exported and analyzed after the procedure. The method was already used during complex catheter ablation as part of a small observational study, but does not yet count as standard monitoring.

So far, it is unclear to what extent a continuous, transcutaneous CO2 monitoring can prevent sedation-associated complications. The aim of this research project is the prospective, randomized analysis of the benefits of continuous, transcutaneous CO2 monitoring + standard monitoring in comparison to the previous standard monitoring. In particular, it should be investigated to what extent sedation-associated complications, such as oxygen saturation decreases, hypercapnia and respiratory acidosis can be prevented by continuous, transcutaneous CO2 monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18 years
2. Indication of electrophysiological intervention with the need for sedation during electrophysiological intervention
3. Written consent

Exclusion Criteria:

1. Lack of written consent of the patient or lack of consent
2. Contraindications / Incompatibilities to the attachment of the adhesive electrode (forehead)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Alteration of oxygen saturation | during procedure
  Oxygen saturation change (spO2 < 90%)
Alteration of pCO2 | during procedure
  pCO2 change of > 30% of the initial value (measured in mmHg)
Hypercapnia | during procedure
  pCO2 > 70 mmHg in the venous blood gas analysis
Respiratory acidosis | during procedure
  pH < 7.25 (respiratory acidosis)

SECONDARY OUTCOMES:
Alteration of systolic blood pressure | during procedure
  systolic blood pressure < 80 mmHg
Alteration of mean blood pressure | during procedure
  mean arterial blood pressure < 65 mmHg
Oxygen saturation change | during procedure
  spO2 < 90%
Change of pCO2 | during procedure
  pCO2 change of > 30% of the initial value (measured in mmHg)
Increase of pCO2 | during procedure
  pCO2 > 70 mmHg in the venous blood gas analysis
Alteraiont of blood pH | during procedure
  pH < 7.25 (respiratory acidosis)
Wake up behaviour | up to 15 minutes postprocedural
  time until the patients is awakened (measured in minutes)
Sedation associated postprocedural complications | up to 30 minutes postprocedural
  postoperative nausea and vomiting (PONV)/Shivering

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Weinmann, PD Dr., Principal Investigator — University of Ulm
Locations (1):
- Ulm University Medical Center, Internal Medicine II, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teumer Y, Buss A, Diofano F, Aktolga D, Katov L, Bothner C, Dahme T, Ochsner W, Mayer B, Rottbauer W, Weinmann-Emhardt K. Prospective randomized evaluation of transcutaneous carbon dioxide monitoring during complex electrophysiological procedures under deep sedation: the TRACES trial. Clin Res Cardiol. 2024 Nov 7. doi: 10.1007/s00392-024-02570-8. Online ahead of print. PMID 39508888